CLINICAL TRIAL: NCT06595277
Title: Study of Clinical Practices for the Management of Neuromuscular Blocking Agents in Cardiac Surgery
Brief Title: Neuromuscular Blocking Agents in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SRB2024216
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Surgery; Neuromuscular Blocking Agents
Keywords: cardiac surgery; neuromuscular transmission; neuromuscular blocking agents
MeSH Terms: interventions — Muscle Relaxation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac surgery with NMBA: All patients undergoing cardiac surgery at Hôpital Érasme between October 1, 2024 and May 31, 2025 who receive any neuromuscular blocking agent.
  Interventions: Diagnostic Test: Neuromuscular blockade

INTERVENTIONS:
Diagnostic Test: Neuromuscular blockade — Neuromuscular blockade will be measured in all patients using a quantitative measurement (TOFScan, IdMed, Marseille, France) during surgery and after surgery until either full neuromuscular recovery or time of scheduled extubation.

SUMMARY:
1. Background:

   Neuromuscular blocking agents (NMBA) are commonly used in cardiac surgery anesthesia to facilitate airway management and ventilation, and ensure optimal operative conditions. To improve post-operative results and reduce the length of stay in the intensive care unit, the concept of "Fast track anesthesia" is coming into force, which includes all techniques that offer extubation within 1-6 hours post-operatively. Fast-track cardiac surgery is only feasible when short-acting NMBA are used and neuromuscular transmission has returned to normal by the end of the operation or just before extubation, a few hours after surgery. This requires quantitative monitoring of muscle strength, the only way to eliminate residual paralysis defined by a TOF ratio ≥ 0.9. The American Society of Anesthesiologists (ASA) and the European Society of Anesthesiology and Intensive Care (EASIC) recommend quantitative measurement of neuromuscular block until extubation.This is the only way to avoid the complications of residual paralysis, essentially postoperative pulmonary complications. The POPULAR study clearly highlighted the shortcomings of current NMBA management: out of a total population of 17150 patients, only 16.5% were extubated, with a TOF ratio greater than 0.90. Cardiac surgery patients are brought to the ICU still sedated, intubated and ventilated. Neuromuscular blocking agents are usually discontinued at the end of surgery. As awakening and extubation take place later in the ICU, clinicians often consider that the action of neuromuscular blocking agents is over, but without making a quantitative measurement as recommended by the guidelines.
2. Objectives of the clinical research project:

   2.1 Primary objective: The primary objective of this single-center prospective observational study is to systematically monitor the degree of postoperative curarization up to the time of extubation, and to assess the degree of adherence of intensive care teams to extubation recommendations based on quantitative measurements of the degree of neuromuscular junction block.

   2.2 Secondary objectives: Quantify NMBA doses used, duration of action, duration of recovery.
3. Methodology of the clinical research project:

   In this study, we will systematically check the degree of curarization of cardiac surgery patients up to the time of extubation. Prior to surgery, all patients will have an explanation of the protocol and will give written informed consent for the use of their data. Patient management is at the discretion of the anaesthetist in charge and will not be altered in any way by the protocol. All drugs used will be "standard of care". At the end of the procedure, one of the investigators will stay with the patient in intensive care and measure the degree of neuromuscular blockade with a curameter used as standard in clinical routine at Erasme Hospital (TOFScan, IdMed, Marseille, France). All measurements will be made in accordance with Good clinical research practice (GCRP) in pharmacodynamic studies of neuromuscular blocking agents III. This measurement will be carried out continuously until the patient is extubated or 100% neuromuscular transmission has been recovered. ICU staff in charge of the patient will be blinded to the measurements done by the investigators. Intensive care physicians manage the patient according to the ICU standard of care. If the patient represents a residual curarization at the time of extubation, the investigators will inform the ICU staff in order to avoid endangering the patient.

   No intervention will be made with regard to the anesthesia and post-operative monitoring protocol; all medications and interventions will be considered "standard of care" and will be left to the discretion of the anesthesiologist and ICU team in charge.
4. Design of the clinical research project:

   This is a prospective, observational study.
5. Participants:

All patients undergoing cardiac surgery at Hôpital Érasme between October 1, 2024 and May 31, 2025.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over
* Patients scheduled for cardiac surgery using a neuromuscular blocker
* Written informed consent

Exclusion Criteria:

* Absence of consent
* Minor patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing cardiac surgery at Hôpital Érasme between October 1, 2024 and May 31, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Concordance with current guidelines | 12 hours
  Percentage of patients (%) where neuromuscular management by ICU staff is in concordance with current guidelines for neuromuscular blocking agents.

SECONDARY OUTCOMES:
TOF ratio at scheduled extubation | 12 hours
  The train of four ratio (TOF ratio) will be measured at the time of scheduled extubation and its value recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Schmartz, MD, Principal Investigator — Université Libre de Bruxelles
Locations (1):
- H.U.B - Hôpital Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuchs-Buder T, Brull SJ, Fagerlund MJ, Renew JR, Cammu G, Murphy GS, Warle M, Vested M, Fulesdi B, Nemes R, Columb MO, Damian D, Davis PJ, Iwasaki H, Eriksson LI. Good clinical research practice (GCRP) in pharmacodynamic studies of neuromuscular blocking agents III: The 2023 Geneva revision. Acta Anaesthesiol Scand. 2023 Sep;67(8):994-1017. doi: 10.1111/aas.14279. Epub 2023 Jun 22. PMID 37345870
- [Background] Kirmeier E, Eriksson LI, Lewald H, Jonsson Fagerlund M, Hoeft A, Hollmann M, Meistelman C, Hunter JM, Ulm K, Blobner M; POPULAR Contributors. Post-anaesthesia pulmonary complications after use of muscle relaxants (POPULAR): a multicentre, prospective observational study. Lancet Respir Med. 2019 Feb;7(2):129-140. doi: 10.1016/S2213-2600(18)30294-7. Epub 2018 Sep 14. PMID 30224322
- [Background] Fuchs-Buder T, Romero CS, Lewald H, Lamperti M, Afshari A, Hristovska AM, Schmartz D, Hinkelbein J, Longrois D, Popp M, de Boer HD, Sorbello M, Jankovic R, Kranke P. Peri-operative management of neuromuscular blockade: A guideline from the European Society of Anaesthesiology and Intensive Care. Eur J Anaesthesiol. 2023 Feb 1;40(2):82-94. doi: 10.1097/EJA.0000000000001769. Epub 2022 Nov 15. PMID 36377554
- [Background] Thilen SR, Weigel WA, Todd MM, Dutton RP, Lien CA, Grant SA, Szokol JW, Eriksson LI, Yaster M, Grant MD, Agarkar M, Marbella AM, Blanck JF, Domino KB. 2023 American Society of Anesthesiologists Practice Guidelines for Monitoring and Antagonism of Neuromuscular Blockade: A Report by the American Society of Anesthesiologists Task Force on Neuromuscular Blockade. Anesthesiology. 2023 Jan 1;138(1):13-41. doi: 10.1097/ALN.0000000000004379. PMID 36520073
- [Background] Hemmerling TM, Russo G, Bracco D. Neuromuscular blockade in cardiac surgery: an update for clinicians. Ann Card Anaesth. 2008 Jul-Dec;11(2):80-90. doi: 10.4103/0971-9784.41575. PMID 18603747